CLINICAL TRIAL: NCT01663701
Title: Simplified Severe Sepsis Protocol-2 (SSSP-2): A Randomized Controlled Trial of a Bundled Intervention for Severe Sepsis at the University Teaching Hospital in Zambia
Brief Title: Simplified Severe Sepsis Protocol-2 (SSSP-2) in Zambia
Acronym: SSSP-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSSP-2; R24TW007988 (NIH)
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Sepsis; Severe Sepsis; Tuberculosis
Keywords: Sepsis; Severe sepsis; Tuberculosis; Bundle; Zambia
MeSH Terms: conditions — Sepsis; Tuberculosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (Active Comparator): Patients are managed according to admitting doctors' orders. Blood cultures are drawn in all patients. Antibiotics are specified by the admitting doctors.
  Interventions: Other: Usual care
- Simplified Severe Sepsis Protocol (Experimental): This protocol consists of an early aggressive fluid strategy, early blood cultures and antibiotics, and, when appropriate, blood transfusion and titratable dopamine. Monitoring is based on physical exam findings. Antibiotics are specified by the admitting doctors.
  Interventions: Other: Simplified severe sepsis protocol

INTERVENTIONS:
Other: Simplified severe sepsis protocol — This protocol consists of an early aggressive fluid strategy, and, when appropriate, blood transfusion and titratable dopamine. Monitoring is based on physical exam findings.
  Arms: Simplified Severe Sepsis Protocol
Other: Usual care — Patients are managed according to admitting doctors' orders
  Arms: Usual care

SUMMARY:
This study is a randomized control trial assessing the impact of a simple evidence-based protocol for the treatment severe sepsis with hypotension in Zambia. This is a follow-up study to the Simplified Severe Sepsis Protocol (SSSP) study. The intervention protocol consists of a scheduled fluid regimen, early blood culture and antibiotics, and dopamine and blood transfusion when necessary. It is hypothesized that the protocol will significantly decrease in-hospital mortality in patients with severe sepsis and hypotension.

DETAILED DESCRIPTION:
In recent years, evidence-based protocols of bundled therapies have improved survival of severe sepsis in developed countries. In sub-Saharan Africa, simple therapies such as IV fluids and early antibiotics are frequently under-utilized. Studies of fluid interventions in the region, however, have demonstrated conflicting results. Outcomes in septic patients may be further affected by delays in the diagnosis of tuberculosis-associated severe sepsis.

The aims of this study are (1) To assess the impact on survival of a simple evidence-based protocol for severe sepsis with hypotensionor septic shock, (2) To evaluate the cost of implementation for a simplified severe sepsis protocol, (3) To develop a clinical diagnostic score for identifying tuberculosis in HIV positive patients with severe sepsis, and (4) To assess the performance of the Xpert TB/RIF rapid PCR system and urine lipoarabinomannan assay for diagnosing tuberculosis in HIV positive patients with severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* infection suspected by the treating physician
* 2 or more of the following SIRS criteria:
* - Heart rate >90/min
* Respiratory rate >20/min
* - Temperature ≥ 38° C or < 36° C
* White blood count > 12,000 or < 4,000/µL
* 1 of the following:
* Systolic blood pressure (SBP) ≤ 90 mm Hg
* Mean arterial blood pressure (MAP) ≤ 65 mm Hg

Exclusion Criteria:

* Gastrointestinal bleed in the absence of fever
* Need for immediate surgery
* Respiratory rate greater than 40/min with oxygen saturation less than 90%
* Suspected congestive heart failure exacerbation
* End-stage renal disease
* Raised jugular venous pressure (JVP) at baseline
* Currently incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
In-hospital all cause mortality | During hospitalization, expected average 14 days

SECONDARY OUTCOMES:
28-day all-cause mortality | 28-day
In-hospital all cause mortality adjusted for illness severity | During hospitalization, expected average 14 days
  Adjusted for SAPS3 score
28-day all cause mortality adjusted for baseline illness severity | 28-day
  Adjusted for SAPS3 score
Cumulative adverse events | During hospitalization, expected average 14 days
  A composite outcome consisting of dopamine extravasation, dopamine-associated tissue ischemia or necrosis, iatrogenic pulmonary oedema, and transfusion-related adverse events.
Treatment cost per patient | During hospitalization, expected average 14 days
  A budget impact analysis will determine the cost of treatment per patient using a mix of direct measurements and micro-cost observation.
Antibiotic changed due to culture results | During hospitalization, expected average 14 days
  The proportion of patients whose antibiotic regimen was changed due to information obtained from blood culture results.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin L Andrews, MD, Principal Investigator — Vanderbilt University and University of Zambia
Locations (1):
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Requests for data sharing should be directed to PI. PI will then confer with Zambian co-PI to confirm that data sharing is allowable by Zambian law.

REFERENCES:
- [Derived] Andrews B, Semler MW, Muchemwa L, Kelly P, Lakhi S, Heimburger DC, Mabula C, Bwalya M, Bernard GR. Effect of an Early Resuscitation Protocol on In-hospital Mortality Among Adults With Sepsis and Hypotension: A Randomized Clinical Trial. JAMA. 2017 Oct 3;318(13):1233-1240. doi: 10.1001/jama.2017.10913. PMID 28973227